CLINICAL TRIAL: NCT02633683
Title: A Multicenter Open-Label Extension Study to Evaluate the Efficacy and Safety of HORIZANT (Gabapentin Enacarbil) Extended-Release Tablets in Adolescents Aged 13 to 17 Years Old With Moderate-to-Severe Primary Restless Legs Syndrome
Brief Title: An Extension Study to Evaluate the Efficacy and Safety of HORIZANT in Adolescents With Moderate-to-Severe Primary RLS
Acronym: RLS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XP110
Record Dates: First submitted 2015-12-10; First posted 2015-12-17 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: RLS
Keywords: Restless Legs Syndrome; RLS
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HORIZANT 600 mg (Experimental): HORIZANT 600 mg once daily
  Interventions: Drug: HORIZANT 600 mg

INTERVENTIONS:
Drug: HORIZANT 600 mg — HORIZANT 600 mg once daily
  Other Names: Gabapentin Enacarbil Extended-Release Tablets

SUMMARY:
The objectives of the trial are to evaluate the long-term efficacy and safety of HORIZANT (Gabapentin Enacarbil) 600 mg daily, for the treatment of RLS in adolescents (13 to 17 years of age) diagnosed with moderate-to-severe primary RLS.

DETAILED DESCRIPTION:
Patients who complete the 12-week daily dosing efficacy and safety study (XP109) will be allowed to enroll in the open-label extension (OLE) study (XP110), thereby providing exposure to HORIZANT for up to 48 weeks. Enrolled patients will take open-label HORIZANT 600 mg tablets once a day at approximately 5 PM with food, beginning at Week 0 of the OLE study up to and including Week 36. After the end of the treatment period, a follow-up visit will be included 14 days (± 3 days) after the last dose of HORIZANT. Patients will visit the clinical site on 6 different occasions, including a follow-up visit 14 days (± 3 days) after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

Patients who completed participation in HORIZANT Study XP109.

* Negative pregnancy test for females of childbearing potential. Male patients able to father a child must agree to use a barrier method (male condom, female condom, diaphragm, or cervical cap) with spermicide for at least 30 days prior to dosing and throughout the study. Fertile, sexually active patients must agree to use 2 medically accepted methods of contraception
* Patients must be willing to refrain from using any drugs that are likely to affect RLS or sleep assessments for the duration of the study.
* Signed patient and parent (or legal guardian) Institutional Review Board (IRB)-approved assent and consent forms before any study procedures are carried out

Exclusion Criteria:

* Patients who, in the opinion of the investigator, would be noncompliant with the study visit schedule, procedures, or medication administration
* Patients who have developed clinically significant or unstable medical conditions, or who would otherwise be unsuitable for participation in a continuation study with gabapentin enacarbil

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression of Improvement (CGI-I) score | Week 12
  assessment at designated timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Steven Caras, MD, Study Director — Xenoport/Arbor Pharmaceuticals, LLC
Locations (11):
- United States (11):
  - Stanford Sleep Medicine Center, Redwood City, California
  - Pacific Research Network, San Diego, California
  - NW FL Clinical Research Group, Gulf Breeze, Florida
  - Florida Pediatric Research Institute, Winter Park, Florida
  - Clinical Integrative Research Center of Atlanta, INC, Atlanta, Georgia
  - Josephson Wallack Munshower Neurology, PC, Indianapolis, Indiana
  - Dent Neurologic Institute, Amherst, New York
  - Mercy Health - Children's Hospital Pulmonary & Sleep Center, Toledo, Ohio
  - The Sleep Center at the Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - SleepMed of South Carolina; SleepMed, Inc., Columbia, South Carolina
  - Vanderbilt University School of Medicine, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No